CLINICAL TRIAL: NCT05618509
Title: Immediate Effects of STENDO on the Walking Abilities of Patients with COPD
Brief Title: Immediate Effects of STENDO on the Walking Abilities of Patients with COPD (STENDO-COPD)
Acronym: STENDO-COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-A01932-39
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: COPD; Walking Performance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient with STENDO (Active Comparator)
  Interventions: Device: STENDO session; Other: A six-minute walking distance test; Other: Near Infrared Spectroscopy
- Patient with placebo (Placebo Comparator)
  Interventions: Other: A six-minute walking distance test; Other: Near Infrared Spectroscopy; Device: STENDO placebo

INTERVENTIONS:
Device: STENDO session — It is a combination enveloping the lower limbs up to the abdomen. The massage system induces pressure from the ankles to the abdomen between each heartbeat. The capacity for physical exercise is potentially improved.
  STENDO : 45 minutes, 2 legs and the pelvis, pression of 65mm Hg
  Arms: Patient with STENDO
Other: A six-minute walking distance test — Before and after STENDO session, the patient has to walk 6 minutes in a flat corridor (30m long)
Other: Near Infrared Spectroscopy — The goal is to measure the evolution of the oxygen consumption of the right leg during an effort on a bicycle at constant power for 5 minutes.
Device: STENDO placebo — STENDO placebo : 45 minutes, on 2 legs and the pelvis, pression of 10 mmHg
  Arms: Patient with placebo

SUMMARY:
The STENDO process is a heart rate synchronized massage system initially validated for the treatment of lymphedema. It is a combination enveloping the lower limbs up to the abdomen. The massage system induces pressure from the ankles to the abdomen between each heartbeat. This technique would also allow an improvement of endothelial function by a greater release of nitric oxide. Thus the capacity for physical exercise is potentially improved.

The use of STENDO has never been evaluated in COPD (Chronic obstructive pulmonary disease) where physical capacity is impaired with, in particular, the presence of endothelial dysfunction. STENDO may improve walking performance. If these hypotheses are validated, the STENDO could be positioned as a complement to the exercise rehabilitation strategies offered to symptomatic COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic chronic obstructive pulmonary disease (COPD) attested by a Tiffeneau ratio <70%
* Not oxygen dependent
* Oriented for an ambulatory effort rehabilitation program in after-care and rehabilitation
* Negative urine pregnancy test in women of childbearing age
* Affiliation to a social security scheme or beneficiary of such a scheme
* Patient having signed the free and informed consent

Exclusion Criteria:

* Neurological or osteo-articular pathology impeding walking.
* Dementia with MMSE (Mini mental state examination) <24/30
* Heart failure
* Covid + in the previous 3 months
* Major surgery in the year preceding the session
* Heavy abdominal, pelvic and lower limb cosmetic surgery in the year preceding the session
* Impaired comprehension and/or expression
* Being simultaneously on oral contraception (pill) and smoking (more than 10 cigarettes per day)
* Severe unbalanced high blood pressure
* severe peripheral neuropathy
* Colostomy
* Open fracture, bleeding or healing wound
* 3rd degree burn
* Liver cirrhosis
* Bedsore
* Have prohibitions and restrictions with a history of phlebitis or recent progressive venous thrombosis (less than 6 months) or arterial disease of the lower limbs stage 3 and 4
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Variation in the 6-minute walk test distance after the performance of the STENDO/STENDO Placebo session compared to the value of the initial 6-minute walk test.. | Baseline to immediately after STENDO/STENDO Placebo procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Polyclinique de l'Ormeau, Tarbes, France

IPD SHARING:
Plan to Share IPD: No